CLINICAL TRIAL: NCT04456179
Title: Evaluation of Sensifree's PPG Based Continuous & Non-Invasive Blood Pressure Monitoring System in Comparison to Invasive Radial Arterial Line
Brief Title: Continuous Non-Invasive Blood Pressure System Data Collection in Comparison to Invasive Radial Arterial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensifree Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR2020-363
Record Dates: First submitted 2020-06-03; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Blood Pressure Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: GE Datex-Ohmeda Oxy-F Finger Clip Pulse Oximeter Sensor — PPG based, fingertip mounted sensor, that measures the oxygen level (oxygen saturation) of the blood and generates a waveform
Device: Arrow® arterial catheterization kit (Teleflex) — Invasive monitoring of blood pressure via catheterization of the radial artery, displaying a continuous pressure waveform

SUMMARY:
The purpose of this study is to evaluate methods to modify blood pressure in humans and measure the effectiveness of such methods. A secondary outcome is to evaluate the performance of an investigational continuous non-invasive blood pressure (cNIBP) device created by Sensifree. The tests will per performed in non-hospitalized subjects under varied controlled conditions that include resting blood pressure and non-pharmacologically induced blood pressure changes.

DETAILED DESCRIPTION:
On a first visit a screening procedure to verify inclusion / exclusion criteria are met will be conducted. On the primary procedure visit, data collection will begin with the subjects having the investigational device, ECG sensors, and 1 or more pulse oximetry sensors placed on them for data collection and to monitor their safety for the duration of the study. A physician will place an arterial line in the radial artery. The Sensifree cNIBP system will be calibrated with an oscillometric and/or auscultatory blood pressure cuff measurement taken on the arm opposite the arterial line.

A series of blood pressure changes will be induced, including various combinations of methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject must be willing and able to comply with study procedures and duration

Exclusion Criteria:

* Subject with a BMI over 39
* Deformities or abnormalities that may prevent proper application of the device under test
* Lateral difference in blood pressure greater than 5mmHg diastolic and 9mmHg systolic
* Tachycardia or resting heart rate less than 45 bpm
* Females who are pregnant, who are trying to get pregnant, (confirmed by positive urine pregnancy test unless the subject is known to be not of child-bearing potential)
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * have had cardiovascular surgery
  * have cardiac pacemakers and/or automatic internal cardio-defibrillator
  * Chest pain (angina)
  * Abnormal pulse pressure
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
  * Pulsus Paradoxus
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with a contact allergy to ultrasound gel.
* Subjects with prior or known allergies to iodine or lidocaine (or similar pharmacological agents, e.g. Novocaine)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test
* Subject is intoxicated during the time of the visit, or was intoxicated within 24 hours prior to study visit, as reported by the subject, or per study staff judgment.
* Other known health condition, should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — At least 30% of the subjects will be female and at least 30% will be male
Enrollment: 6 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the magnitude of blood pressure change (measured in mmHg) cause by different isometric efforts in humans | 3-4 hours per subject
  Measure the effect of a combination of the following isometric efforts on a subject's blood pressure (measured in mmHg):
  1. Hand grip
  2. Weight lifting
  3. Leg static effort

SECONDARY OUTCOMES:
Measure the accuracy of an investigational continuous non-invasive blood pressure (cNIBP) device | 3-4 hours per subject
  Comparison of BP values (Systolic, Diastolic, MAP) that are calculated by the investigational device to the BP values measured by the arterial line during isometric effort comprising a combination of the following isometric efforts on a subject's blood pressure:
  1. Hand grip
  2. Weight lifting
  3. Leg static effort

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Ruiz Cabrera, M.D, Principal Investigator
Locations (1):
- Clinimark Lab, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No